CLINICAL TRIAL: NCT06750198
Title: Effects of Hip Focused Exercises on Pain, Range of Motion, Functional Disability, Muscle Strength and Endurance in Patients With Post Operative Anterior Cruciate Ligament Rehabilitation
Brief Title: Effects of Hip Focused Exercises in Patients With Post Operative Anterior Cruciate Ligament Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0109
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Anterior Cruciate Ligament Rehabilitation
Keywords: Anterior cruciate ligament Rehabilitation; Hip focused Exercises; pain; Range of Motion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip focused exercises (Experimental): will receive hip focused exercises and standard rehabilitation protocol with the frequency of 2 sets and 10 repetitions thrice per week for a total of 12 weeks. Pre and post intervention values will be taken on 1st day and after 12 weeks.
  Interventions: Other: Hip focused; Other: Standard rehabilitation
- Standerd rehab protocol (Active Comparator): will receive only standard rehabilitation protocol with the frequency of 2 sets and 10 repetitions thrice per week for a total of 12 weeks. Pre and post intervention values will be taken on 1st day and after 12 weeks
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Hip focused — Group A will be treated with hip focused exercises and standard rehabilitation protocol.
  Hip focused exercises will be comprised of following exercises in phase 1 will be Side lying hip abduction, Hip abduction in standing, Hip extension from prone, Single leg bridge, Side lying clam with resistance while exercises in phase 2 will be same with more repetitions in addition to Side lunges, Forward lunges
  Arms: Hip focused exercises
Other: Standard rehabilitation — Group B will be only be treated with standard rehabilitation protocol. When participant reach full ROM of knee, perform four sets of 20 repetitions of straight leg raising with full extension, and maintain one minute single leg balance on a solid surface with the affected side, subject can transfer to phase 2

SUMMARY:
A Randomized Controlled Trial will be conducted at Mahaban Medical and Research Hospital through consecutive sampling technique on 66 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with hip focused exercises and standard rehabilitation protocol while Group B will be treated with traditional exercises at the frequency of 2 sets with 10 repetitions and thrice a week. Outcome measures will be conducted through pain, range of motion, functional disability, muscle strength and endurance after 12 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non- parametric test will be used within a group or between two groups.

DETAILED DESCRIPTION:
Anterior cruciate ligament plays an important role in knee stability and is prone to contact and and non-contact injuries. ACL reconstruction followed by proper rehabilitation is the most successful procedure to restore knee stability and ROM. Keeping in mind the lower limb kinematics and biomechanics the aim of this study will be to see the effects of hip focused exercises on pain, range of motion, functional disability, muscle strength and endurance in patients with post-operative ACL rehabilitation. A Randomized Controlled Trial will be conducted at Mahaban Medical and Research Hospital through consecutive sampling technique on 66 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with hip focused exercises and standard rehabilitation protocol while Group B will be treated with traditional exercises at the frequency of 2 sets with 10 repetitions and thrice a week. Outcome measures will be conducted through pain, range of motion, functional disability, muscle strength and endurance after 12 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non- parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

Both males and females of age group between 18 and 45 years

* Patients with ACL reconstruction in early rehabilitation phase.
* Physically or recreationally active a minimum of three times per week.(26)
* 1-5 day post operatively(26)
* Physically healthy and without patients with other medical history or joint deformities
* Patients without severe meniscus or cartilage damage (27)
* Complaints of pain (NPRS 3-7) and swelling in the operated knee

Exclusion Criteria:

Patients with multiple ligament injuries in the knee joint

* Patients with knee osteoarthritis
* Patients with joint infection (27)
* An associated chondral defect requiring surgical intervention
* A meniscus tear requiring a repair.
* Patients with incomplete follow-up (28)
* Presence of unstable medical conditions preventing the patient from participating in the rehabilitation program.
* History of ipsi-lateral hip replacement
* Ipsi-lateral hip osteoarthritis or lateral hip pain
* Neurological or any other conditions affecting strength or function of lower limbs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale (NPRS) | 6 WEEK
  The Numeric Pain Rating Scale (NPRS) is commonly used in the clinical setting and is convenient to administer and interpret. The NPRS is a numbered scale that begins with zero and ends at ten. Zero indicates no pain, while ten is the worst intensity of pain that individual can imagine
Universal Goniometer | 6th week
  The goniometer is used to objectively assess active and passive joint ROM. The universal or standard plastic, long armed, 360 degree goniometer is frequently recommended for measurement of knee ROM as the longer arm is thought to reduce error resulting from incorrect placement of the goniometric axis
WOMAC | 6th week
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used to measure the physical function of the knee. This scale was shown to be a valid and reliable tool, which was utilized to assess the physical function in patients with knee surgery. This tool comprises 24 questions: 5 questions about pain (0-20 points), 2 questions about stiffness (0-8 points), and 17 questions about physical functions difficulty (0-68 points), which may be completed in less than 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsumoto H, Suda Y, Otani T, Niki Y, Seedhom BB, Fujikawa K. Roles of the anterior cruciate ligament and the medial collateral ligament in preventing valgus instability. J Orthop Sci. 2001;6(1):28-32. doi: 10.1007/s007760170021. PMID 11289582
- [Background] Petersen W, Tillmann B. Structure and vascularization of the cruciate ligaments of the human knee joint. Anat Embryol (Berl). 1999 Sep;200(3):325-34. doi: 10.1007/s004290050283. PMID 10463347
- [Background] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430